CLINICAL TRIAL: NCT05842720
Title: Consented Unsedated Endoscopy in High Risk Patients That Require Anesthesiologist Observation During the Procedure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-7848-20-ML-CTIL
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- retrospective (Active Comparator): Consecutive patients with ASA score≥3 that underwent unsedated colonoscopy from May 2021 to August 2022 at Sheba medical center were identified by search of the computerized endoscopy database). Following an informed consent, patients were interviewed over the phone using a structured questionnaire. To assess their satisfaction, a standard Likert scale between 1 (unsatisfied) to 5 (very satisfied) was administered. Additional assessment included the maximum level of pain experienced at any point during the procedure (between 1-no pain) to 5-severe pain), and whether they would choose to perform future procedures without sedation in the future. Patients were also asked if they were able to return on the same day to their routine daily function and activities
  Interventions: Procedure: un-sedated colonoscopies
- prospective (Active Comparator): High risk patients scheduled for an anesthesiologist-assisted sedated-colonoscopy in Sheba medical center, were contacted during their clinic visit or by phone to receive explanation about the option to enroll in this unsedated colonoscopy study.
  After obtaining informed consent, patients' Anxiety trait was assessed with the help of State-Trait Anxiety Inventory (STAI) questionnaire [8] in order to assess their level of anxiety and to investigate its predictive utility for their success in undergoing the unsedated procedure. Upon completion of the procedure in the same satisfaction questionnaire was administered, as detailed above for the retrospective part
  Interventions: Procedure: un-sedated colonoscopies

INTERVENTIONS:
Procedure: un-sedated colonoscopies — un-sedated colonoscopies in high risk patients with ASA>=3

SUMMARY:
This study aim to examine the safety and feasibility of unsedated colonoscopy in patients with high risk for sedation (ASA score≥3).

DETAILED DESCRIPTION:
This was a two-part study: Part 1 was a retrospective study of patients with ASA score≥3 that underwent unsedated colonoscopy from May 2021 to August 2022 at Sheba medical center, who were contacted up to one year after the procedure and were asked to assess their satisfaction and pain level on a standard Likert score from 1-5. Part 2 was a prospective study which included high risk patients who were scheduled for an anesthesiologist-assisted sedated-colonoscopy and who consented to undergo an unsedated procedure. The primary outcome was patients' satisfaction during and up to one week after the procedure. Pain level, adverse events and hemodynamic parameters during the procedure were secondary outcomes. Baseline State-Trait Anxiety Inventory (STAI) questionnaire were also administered and results examined vis-à-vis satisfaction scores

ELIGIBILITY:
Inclusion Criteria:

* Only adults (>18 years of age) that will be assessed as high risk and require an anesthesiologist clinic assessment prior to the procedure and anesthesiologist presence during the procedure.

Exclusion Criteria:

1. Patients that are planned to go through both gastroscopy and colonoscopy procedures.
2. Patients with known adhesions and/or prior small bowel obstructions.
3. Patients that are planned to have a complicated procedure (complicated polypectomy etc).
4. Patients that are not able to give their consent with a full understanding of the procedure.
5. Patients that are pregnant.
6. Patients with a heart rate above 120 bpm or less than 40 bpm at the baseline as measured before starting the procedure.
7. Patients with a systolic blood pressure above 180mmHg or bellow 90mmHg as measured at the baseline before starting the procedure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
satisfaction rate | up to 1 week after the date of the procedure
  Overall satisfaction score as assessed by Likert scale post-procedure

SECONDARY OUTCOMES:
Recovery time after the procedure | up to 24 hours after the procedure
  the time lapse between extraction of colonoscope from the rectum and discharge of the patient from the Endoscopy recovery unit.
Complications or adverse effects rates during the procedure | from the beginning of the procedure until the end of the procedure
  perforations, post-polypectomy bleeding, bradycardia (defined as pulse rate under 40 bpm), low oxygen saturation (defined as saturation below 90% under nasal oxygen cannula) or hemodynamically instability (defined as systolic blood pressure below 90mmHg and diastolic blood pressure below 60mmHg)
Complete examination rates | from the beginning of the procedure until the end of the procedure
  how many examination were completed up to cecum intubation without need for sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center Tel Hashomer, Ramat Gan, Israel